CLINICAL TRIAL: NCT03503721
Title: Bipolar Transurethral Enucleation (BipolEP) vs Bipolar Transurethral Resection of the Prostate: A Prospective Interventional Multi-center Randomized Controlled Trial
Brief Title: Bipolar Transurethral Enucleation (BipolEP) vs Bipolar Transurethral Resection of the Prostate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Dr. Thomas Kunit, Vice Chairman, Department of Urology and Andrology, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2018-01-17; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Benign Prostatic Hyperplasia; Bladder Outlet Obstruction
Keywords: BipolEP; TURP
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BipolEP (Experimental): includes all patients undergoing BipolEP surgery
  Interventions: Procedure: BipolEP
- TURP (Active Comparator): includes all patients undergoing TURP surgery
  Interventions: Procedure: bipolarTURP

INTERVENTIONS:
Procedure: BipolEP — the prostate will be transurethrally enucleated using a bipolar current
  Arms: BipolEP
Procedure: bipolarTURP — the prostate will transurethrally resected using a bipolar current
  Arms: TURP

SUMMARY:
The aim of this study is to compare two different surgical methods for treating benign prostatic obstruction (BPO).

The investigators are going to compare the risks and benefits of bipolar transurethral resection of the prostate (TURP) and bipolar transurethral enucleation of the prostate (BipolEP). Furthermore, the investigators are going to compare the amount of tissue resected per minute, in order to assess the efficiency of each surgical method.

It is a prospective, interventional, multi-centre (2 centres total), randomized trial.

Approximately 84 patients will be included

DETAILED DESCRIPTION:
Overview:

The aim of this study is to compare two different surgical methods for treating benign prostatic obstruction (BPO).

The investigators are going to compare the risks and benefits of bipolar transurethral resection of the prostate (TURP) and bipolar transurethral enucleation of the prostate (BipolEP). Furthermore, the investigators are going to compare the amount of tissue resected per minute, in order to assess the efficiency of each surgical method.

All patients will be followed up for 12 months. All the examinations used to assess the risks and benefits of BipolEP and TURP are listed below:

* Dysuria visual analogue scale (at 1 month)
* I-PSS (international prostate symptom score), QOL (quality of life), Qmax (maximum flow rate of urine) and PVR (post void residual bladder volume) before surgery and at 1, 4 and 12 months
* IIEF-15 (international index of erectile function) and PSA (prostate specific antigen) (before surgery and at 4 and 12 months)
* TRUS (transrectal ultrasonography) for prostate size before surgery and at 4 months

It is a prospective, interventional, multi-centre (2 centres total), randomized trial.

Approximately 84 patients will be included in this study. Each patient will be randomly assigned either to the BipolEP or to the TURP study arm. For the allocation of treatment to subjects the minimization method will be used (Strata: 1. prostate 60 to 80 ml / more than 80 ml; 2. catheterized / non-catheterized). The minimization procedure will be applied centrally (by the coordinating centre).

Statistical analysis plan :

Concept

The study is designed as a comparison of two kinds of treatment:

Group BipolEP: Bipolar transurethral enucleation of the prostate Group TURP: Bipolar transurethral resection of the prostate

Two primary endpoints are chosen:

1. : IPSS after 12 month [-]
2. : Tissue resection [g/min]

The use of a gate keeping approach makes it unnecessary to adjust the type I error. Primary endpoint (1) will be investigated by a non-inferiority approach (type I error = 5% one-sided), primary endpoint (2) by a superiority approach (type I error = 2.5% one-sided).

Hypotheses:

1. : H-01: Compared to group TURP, IPSS after 12months in group BipolEP is higher (non-inferiority range = 3) H-11: Compared to group TURP, IPSS after 12months in group BipolEP is not higher (non-inferiority range = 3)
2. : H-02: Compared to group TURP, tissue resection in group BipolEP is not increased H-12: Compared to group TURP, tissue resection in group BipolEP is increased

Statistical Methods:

Group Comparisons:

Primary Endpoint (1):

Data (if appropriate, in logarithmised version) will be checked for normal distribution (Kolmogorov-Smirnov with Lilliefors significance correction, type I error = 10%). Hypotheses (H-01, H-11) will be investigated either by a parametric or by a non-parametric one-sided test of equivalence (equivalence range one-sided = 3; type I error = 5% one-sided).

Primary Endpoint (2):

Data (if appropriate, in logarithmised version) will be checked for normal distribution (Kolmogorov-Smirnov with Lilliefors significance correction, type I error = 10%). Hypotheses will be investigated either by the t-test for independent samples or by the Mann-Whitney U-test (type I error = 2.5% one-sided). Hypotheses (H-02, H-12) will be tested only if H-01 hypothesis is rejected.

Further Variables:

All other variables will be analysed by usual parametric and non-parametric tests for univariate comparisons of independent samples.

Two-sided 95% confidence intervals:

For selected variables, two-sided 95% confidence intervals will be calculated.

Type I error adjustment:

No adjustment for the type I error will be made. Therefore - apart from hypotheses testing - the results of inferential statistics will be descriptive only.

Sample size assessment:

The following scenario was used for the sample size estimation concerning primary endpoint (1):

* Non-inferiority range = 3
* Type I error = 5% one-sided
* Type II error = 10%
* IPSS after 12 months in both groups (Mw ± SD) = 4 ± 4
* n (group BipolEP) / n (group TURP) = 1 / 1
* Parametric test The result of the sample size estimation is a requirement of 31 cases per group. Assuming a drop-out rate of 20% and considering the possible need for a non-parametric test a total of 84 inclusions (n=42 / group) are chosen as the sample size of the study.

Data management and quality assurance:

In order to assure that the collected data are accurate, consistent, complete and reliable, the primary investigator will review all the CRFs. If any data is missing, incomplete or inaccurate, the medical record of the patient will be used to identify the missing data. If the data notated in the medical record is missing or implausible, the data will be recorded in the database as missing value. In the intention to treat population and only for the two primary endpoints, the missing values will be replaced according to the worst-case principle (use of the worst assessed value in the study).

After all the CRFs have been checked for completeness and accuracy, the data will be entered in a special database. A second person, involved in the study, will check all the data entered. Once the database is complete and has been checked, it will be locked, marking the beginning of the statistical analysis. The data will be analyzed by a statistician.

The investigator will keep all source documents, CRFs and trial documentation. The investigator will store all study documents and all mandatory documents linked to the study including the identity of all patients (enough information to link the records, eg, the CRF and hospital records), all original signed informed consent forms and copies of all CRD (clinically relevant documents) for a minimum of 5 years. All study-linked documents will be stored under strict security and will be available for review for authorized personnel only.

Adverse Event:

The Investigator and designated study personnel will monitor each subject for adverse events during the study. All adverse events reported between consent and final follow-up will be recorded in the case report form (CRF). The investigator or designee will ask the subject non-leading questions in an effort to detect adverse events. The intra- and postoperative adverse events will be quantified according to the Clavien-Dindo classification. In case of any adverse event or change of treatment, the primary investigator has to be informed.

ELIGIBILITY:
Inclusion Criteria:

* Refractory LUTS (lower urinary tract symptoms) secondary to BPH benign prostate hyperplasia)
* I-PSS greater than 15
* QOL score 3 or greater
* Qmax less than 15 ml per second or patients with acute urinary retention secondary to BPH in whom trial of voiding failed
* Prostate size on preoperative TRUS of 40 to 150 ml

Exclusion Criteria:

* Patients with neurological disorder
* Active urinary tract infection, active bladder or prostate cancer

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-01-18 (Estimated); Study Completion 2021-06-18 (Estimated)

PRIMARY OUTCOMES:
Long-term outcome - Change in IPSS (Difference in IPSS before and 12 months after surgery) | Start: before the surgery End: 356 days after surgery
  The long-term outcome will be measured by comparing the change in IPSS (International Prostate Symptom Score) before and 12 months after surgery. The IPSS is based on the answers to seven questions concerning urinary symptoms (Incomplete emptying, Frequency, Intermittency, Urgency, Weak Stream, Straining, Nocturia) and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic) Question eight refers to the patient's perceived quality of life.

SECONDARY OUTCOMES:
Efficiency of surgical intervention (tissue resected intraoperatively per minute) | Intraoperative
  In order to asses the efficiency of the surgical intervention, the amount of prostate tissue (grams) surgically removed per minute will be recorded. The investigators do want to see whether prostate tissue can be resected faster by using any of the two methods.

OTHER OUTCOMES:
Safety of surgical intervention (comparison of adverse events using the Clavien Dindo-Classification) | Start: start of the surgery End: 356 days after surgery
  All possible adverse events after applying BipolEP or TURP will be assessed using the Clavien-Dindo score. The investigators do want to find out whether the surgery can be performed safer by using BipolEP or TURP.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kunit, MD, Principal Investigator — Vice Chairman
Locations (2):
- Universitätsklinik für Urologie und Andrologie, Salzburger Landeskliniken, Salzburg, Austria
- Urologische Klinik Spital Thurgau, Kantonsspital Frauenfeld, Frauenfeld, Thurgau, Switzerland

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03503721/Prot_SAP_000.pdf